CLINICAL TRIAL: NCT04157257
Title: An Open-Label Phase 2 Study to Evaluate Safety and Efficacy of QL-007 Tablets in Combination With Entecavir or Tenofovir in Patients With Chronic Hepatitis b Who Have Received Nucleoside (Acid) Therapy : a Multicenter, Randomized, Positive Controlled Clinical Trialcontrolled Clinical Trial
Brief Title: An Study to Evaluate Safety and Efficacy of QL-007 Tablets in Combination With Entecavir or Tenofovir in Patients With Chronic Hepatitis b Who Have Received Nucleoside (Acid) Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL-007-202
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis b
Keywords: nucleoside (acid) therapy
MeSH Terms: conditions — Hepatitis B, Chronic; Heartburn | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QL-007 +TDF (Experimental): QL-007 200 mg BID +TDF 300 mg QD
  Interventions: Drug: TDF tablet; Drug: QL-007
- QL-007 +Entecavir (Experimental): QL-007 200 mg BID +Entecavir 0.5 mg QD
  Interventions: Drug: Entecavir Tablet; Drug: QL-007
- TDF monotherapy (Active Comparator): TDF tablet 300 mg QD
  Interventions: Drug: TDF tablet
- Entecavir monotherapy (Active Comparator): Entecavir tablet 0.5 mg QD
  Interventions: Drug: Entecavir Tablet

INTERVENTIONS:
Drug: TDF tablet — TDF tablet 300mg QD
  Other Names: Tenofovir dipirofurate fumarate tablet
  Arms: QL-007 +TDF; TDF monotherapy
Drug: Entecavir Tablet — Entecavir tablet 0.5mg QD
  Other Names: Entecavir
  Arms: Entecavir monotherapy; QL-007 +Entecavir
Drug: QL-007 — QL-007 tablets 200mg BID
  Other Names: QL-007 tablet
  Arms: QL-007 +Entecavir; QL-007 +TDF

SUMMARY:
This is an open label, randomized, multi-center, comparative study. Subjects will be screened prior to study entry to establish eligibility. 60 Subjects who meet all the selection criteria will be randomly assigned to (A) QL007 200mg BID+ Tenofovir dipirofurate fumarate （TDF）300 mg QD, (B) QL007 200 mg BID+ Entecavir 0.5 mg QD, (C)TDF 300 mg QD, (D) Entecavir 0.5 mg QD.

The purpose of this study was to evaluate the efficacy and safety of QL-007 tables in combination with TDF or Entecavir in patients with chronic hepatitis b who have received nucleoside (acid) therapy, and to recommend a reasonable regimen for phase III study.

DETAILED DESCRIPTION:
The subjects received the drug treatment for a maximum of 96 weeks: divided into two stages: the first stage: 0-24 weeks as the core treatment period, 25-48 weeks as the extended treatment period. The second stage: 49-96 weeks is the extended treatment period. Stage 2: subjects in stage 1 group A and C were grouped into group E(QL-007 200 mg BID或XX mg +TDF 300 mg QD), and subjects in group B and D were grouped into group F(QL-007 200 mg BID或XX mg + Entecavir 0.5 mg QD). Subjects in group E and F entered the second stage of treatment according to 200 mg BID. After the efficacy data of the original treatment clinical trial (protocol 201) determine the optimal dose of 007, all subjects entering the second phase will receive the optimal dose of 007 and continue treatment withTDF or Entecavir tablets (007 XXmg+TDF or ETV) into the second phase 49-96 weeks of extended treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years (inclusive) with chronic HBV infection prior to baseline;
2. Subjects who have received a entecavir or tenofovir ester treatment for more than 1 year before screening ;
3. HBsAg > 250 IU/mL and HBV DNA < 60 IU/mL at screening period;
4. ALT≤ 2×ULN;
5. Participants must have understood and signed the ICF.

Exclusion Criteria:

1. Confirmed co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis D virus (HDV);
2. History of liver disease other than chronic hepatitis B;
3. History of Gilbert's Disease;
4. History of decompensated liver disease or any sign of decompensated liver disease at the screening period;
5. Evidence of moderate or severe fibrosis or cirrhosis;
6. Evidence of HCC or AFP > 50 ng/ml at the screening period.
7. Any Clinical laboratory values meet the certain standards at the screening period;
8. Subjects have clinically significant, uncontrolled heart disease and/or recent cardiac event;
9. Risks of serious kidney and respiratory diseases;
10. Impaired gastrointestinal (GI) function or GI disease that may alter absorption of QL-007 as determined by the Investigator;
11. Receiving medications that meet one of the following criteria and that cannot be discontinued ≥1 week prior to the start of treatment QL-007:

    * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes;
    * Moderate or strong inhibitors or strong inducers of CYP3A4
12. Intake of any drugs that can reduce enzyme activity;
13. History of bleeding diathesis;
14. Risks of mental and nervous system diseases during screening;
15. Pregnant or lactating female subjects; Female subjects of childbearing age who were not willing to use effective contraception throughout the study period or male subjects whose partners were fertile but were not willing to use effective contraception;
16. Volunteers who took an Investigational Product within 3 months or who have been within 5 half-lives of other trial drugs before the randomization;
17. Any other condition , which in the opinion of investigator would make a patient unfit for participation in a clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Main index of pharmacodynamics | 24 weeks
  The change of HBsAg levels at week 24 compared to baseline

SECONDARY OUTCOMES:
The secondary pharmacodynamic index | 96 weeks
  The changes of HBsAg and HBeAg level at week 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96 compared to baseline
The secondary pharmacodynamic index | 96 weeks
  The percentage of subjects with HBsAg and HBeAg serological clearance and/or seroconversion at 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96 weeks
The secondary pharmacodynamic index | 96 weeks
  The percentage of subjects with normal ALT level at weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84 and 96
Other evaluation indexes of pharmacodynamics exploration | 96 weeks
  The changes of HBV RNA and HBcrAg compared with baseline at week 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84 and 96
To evaluate the safety of QL-007 in combination with TDF or Entecavir: incidence of adverse events | 96 weeks
  The incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, PhD, Principal Investigator — Southern Hospital of Southern Medical University; Junqi Niu, PhD, Principal Investigator — The First Hospital of Jilin University
Locations (2):
- China (2):
  - Southern Hospital of Southern Medical University, Guangzhou, Guangdong
  - The first hospital of jilin university, Changchun, Jilin